CLINICAL TRIAL: NCT02370550
Title: Cyclosporine A in the TReatment of Interstitial Pneumonitis Associated With Sjogren's Syndrome(CTRIPS): A Prospective, Randomized, Multicenter, Double-Blind Placebo-Controlled Trial
Brief Title: Cyclosporine A in the TReatment of Interstitial Pneumonitis Associated With Sjogren's Syndrome
Acronym: CTRIPS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Zhanguo Li, Professor of Medicine, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2014-M03; U1111-1167-1974 (Other: WHO ICTRP); ChiCTR-IPR-15005990 (Registry Identifier: Chinese Clinical Trial Registry)
Record Dates: First submitted 2015-02-18; First posted 2015-02-25 (Estimated); Last update posted 2020-05-22 (Actual); Status verified 2020-05

CONDITIONS: Sjogren's Syndrome
MeSH Terms: conditions — Sjogren's Syndrome | interventions — Cyclosporine; Long-Term Synaptic Depression; Prednisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cyclosporin A(CsA)+glucocorticoid (Experimental): A. The efficacy/safety are evaluated at V3, V4, V5 and V6, and the treatment is adjusted accordingly. Patients who experienced treatment failure (FVC absolute decrease >15% of predicted values after 4 weeks of treatment) are suggested to switch to intravenous glucocorticoid + cyclophosphamide(CYC) 0.5-1 g/m2 every 4 weeks as the rescue therapy after unblinding, and continue to complete the subsequent follow-up. Each patient can only have one chance to be rescued. Patients who experience a second treatment failure should be withdrawn from the trial and be given empirical treatment. Patients who did not experience treatment failure continued to receive current treatment. B. For subjects with aggravated shortness of breath and dyspnea in between of two consecutive visits, the investigators should decide whether a visit should be increased to complete subsequent examinations.
  Interventions: Drug: Cyclosporin A; Drug: Prednisone; Drug: Calcium carbonate D
- placebo+glucocorticoid (Placebo Comparator): A. The efficacy/safety are evaluated at V3, V4, V5 and V6, and the treatment is adjusted accordingly. Patients who experienced treatment failure are suggested to switch to glucocorticoid + CsA 2-3mg/kg/d, BID as the rescue therapy, and continue to complete the subsequent follow-up. Each patient can only have one chance to be rescued. Patients who did not experience treatment failure continued to receive current treatment. B. For subjects with aggravated shortness of breath and dyspnea in between of two consecutive visits, the investigators in each center should decide whether a visit should be increased.
  Interventions: Drug: Prednisone; Drug: Placebo; Drug: Calcium carbonate D

INTERVENTIONS:
Drug: Cyclosporin A — CsA 2-3 mg/kg/d, BID PO
  Other Names: Cyclosporin A Capsules, CsA soft capsules 25 mg, Hangzhou China-US East China pharmaceutical Co., Ltd.
  Arms: Cyclosporin A(CsA)+glucocorticoid
Drug: Prednisone — Prednisone 0.5mg/kg/d QD PO starting at Week 0. After 2-4 weeks, the initial dose is gradually tapered by 2.5 mg each week until a maintenance dosage of 5-7.5 mg/d through week 52 (visit 6). The initial and maintenance doses are determined by the investigators of each center depending on the patients.
Drug: Placebo — Placebo tablet 2-3 mg/kg/d, BID PO
  Arms: placebo+glucocorticoid
Drug: Calcium carbonate D — Calcium carbonate D 600 mg, QD PO

SUMMARY:
The purpose of this large multicenter, randomized, double-blinded, controlled clinical study is to investigate the efficacy and safety of Cyclosporin A for primary Sjogren's syndrome associated pneumonitis(pSS-IP), which has important implications for the establishment of standardized diagnosis and treatment of pSS-IP.

ELIGIBILITY:
Inclusion Criteria:

* Patients meeting the 2002 or 2012 pSS criteria;
* Patients meeting the diagnostic criteria of interstitial pneumonitis(IP);
* Patients with exertional dyspnea consistent with grade 2 on the Magnitude of Task component of the Mahler Modified Dyspnea Index;
* Pulmonary function test: patients with percentages of forced vital capacity (FVC) to predicted values≥45%, percentage of diffusing capacity of carbon monoxide (DLco) to predicted values≥30%, forced expiratory volume in one second (FEV1) / FVC> 65%;
* For patients who received oral glucocorticoid, the doses should be no more than 10 mg/d (or equivalent amount of other types of glucocorticoids);
* Patients who had not received any prior treatment with immunosuppressants (including but not limited to CYC, CsA, azathioprine(AZA), tacrolimus(FK-506), methotrexate, leflunomide, etc.) or had discontinued the therapy above for at least 3 months; for patients who received hydrochloroquine(HCQ), the doses should be stabilized for at least 3 months;
* Patients who had not received any prior treatment with biological agents, including but not limited to rituximab, infliximab, adalimumab, etanercept, etc., or had discontinued therapy for at least three months;
* For patients who had prior treatment with N-acetylcysteine, the doses of above drugs should be stabilized for at least 3 months;
* The women of reproductive age who had a negative urine pregnancy test. The women and men of reproductive age must receive effective contraceptive measures from the screening period to last administration of drugs;
* Patients who were able to read, to understand and to sign informed consent.

Exclusion Criteria: Patients who met any of the following criteria will not participate in this study.

* Patients with acute exacerbation of IP(AEIP);
* Arterial blood gas analysis showed respiratory failure;
* Patients with lung diseases other than IP:

  1. Patients with severe pulmonary hypertension who require specific treatments assessed by the rheumatology and immunology experts in various clinical centers;
  2. Patients with a history of smoking within the last 6 months or current smokers;
  3. Patients with other serious lung diseases, such as lung tumor or active pulmonary infection;
  4. Lung biopsy, alveolar lavage or high-resolution computerized tomography (HRCT) suggested serious lung diseases other than IP;
* Patients with other rheumatic autoimmune diseases, including but not limited to rheumatoid arthritis, systemic lupus erythematosus, inflammatory myopathy, systemic sclerosis, primary biliary cirrhosis, etc.;
* Patients with serious heart, liver, kidney diseases, hematologic and/ or endocrine diseases:

  1. Heart diseases: decompensated heart failure or refractory hypertension; clinically important abnormal ECG that may lead to unacceptable risks to enrolled patients at screening;
  2. Liver function: alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) ≥2 times the upper limit of normal (ULN);
  3. Renal function: renal tubular and/or interstitial diseases, renal insufficiency: serum creatinine≥2 ULN or glomerular filtration rate (eGFR) <90 ml/min/1.73 m2;
  4. White blood cell (WBC) count <3 ×109/L and/or hemoglobin (Hb) <100 g/L and/or platelet (PLT) count <80×109 /L;
  5. Other serious diseases: such as cancer, etc.;
* Patients with active infection or other diseases which will be aggravated with treatment of glucocorticoid and immunosuppressive therapy;
* Patients positive for HBsAg or hepatitis C antibody;
* Women during pregnancy or lactation, or cannot guarantee effective contraception;
* Patients who did not cooperate with treatment for mental illness or other reasons;
* Patients who had allergic constitution or were allergic to many drugs;
* Patients who were allergic or intolerant to CsA, CYC, or glucocorticoid.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2015-03 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
The forced vital capacity (FVC) | the 52 weeks
  The FVC is expressed as percent of expected values corrected baseline level.

SECONDARY OUTCOMES:
The diffusing capacity of carbon monoxide (DLco) | the 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Zhanguo Li, MD, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China